CLINICAL TRIAL: NCT00766246
Title: A Multicenter, Open-Label, Randomized, Phase II Trial of Docetaxel, Carboplatin and Bevacizumab as First-Line Treatment, Followed by Bevacizumab Plus Pemetrexed Versus Pemetrexed Alone as Second-Line Treatment of Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Phase II Avastin Trial for Stage IIIB/IV NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding support
Sponsor: Pharmatech (Industry)
Collaborators: Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-009; NCT00735891 (obsolete NCT alias)
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV
Keywords: Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First-line (Experimental): Carboplatin, docetaxel, bevacizumab Open-label, single arm with treatment period up to 6 cycles. Patients completing a total of 2 to 6 cycles of first-line without disease progression will be eligible for maintenance.
  Interventions: Drug: bevacizumab; Drug: docetaxel; Drug: carboplatin
- Maintenance (Experimental): Bevacizumab Open-label, single arm with treatment period up to 18 cycles.
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — 15 mg/kg administered in 21 day cycles on day 1 of each cycle for first-line and maintenance
  Other Names: Avastin
Drug: docetaxel — 75 mg/m2 administered in 21-day cycles on day 1 of each cycle for first line treatment
  Other Names: Taxotere
  Arms: First-line
Drug: carboplatin — AUC=6 administered in 21-day cycles on day 1 of each cycle for first-line treatment
  Other Names: Paraplatin
  Arms: First-line

SUMMARY:
This is a randomized, open-label, multicenter study in 160 patients in first line treatment and 114 in second line treatment with advanced or metastatic NSCLC (Stage IIIB/IV).

DETAILED DESCRIPTION:
This phase II clinical trial will address the issues of bevacizumab treatment duration and treatment safety as first-line therapy for patients with non-squamous NSCLC. Following disease progression or treatment failure, the potential benefit of continued bevacizumab therapy will be tested by randomizing patients to two treatment arms, including second-line chemotherapy with or without further bevacizumab. It is hypothesized that continuation of bevacizumab with pemetrexed as second-line treatment following progression will result in improved clinical outcomes for patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed stage IIIB with malignant pleural effusion or stage IV NSCLC except squamous-cell carcinoma
* Measurable disease defined by RECIST
* Adequate organ function:

  1. Absolute neutrophil count ≥ 1.5 x 10(9)/L
  2. Hemoglobin ≥ 9.0 g/dL
  3. Platelets ≥ 100 x 10(9)/L
  4. Hepatic enzyme levels: AST and ALT and Alkaline Phosphatase must be within range allowing for eligibility. In determining eligibility, the more abnormal of the two values (AST or ALT) should be used according to table listed in the protocol
  5. Bilirubin ≤ ULN
  6. Serum Creatinine ≤ 1.5 mg/dL (or creatinine clearance ≥ 60mL/min)
  7. Urine protein/creatinine ratio < 1.0 OR urine dipstick for proteinuria < 2 + (patients discovered to have ≥ 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤1g of protein in 24 hours to be eligible)
  8. INR ≤ 1.5
  9. PTT ≤ ULN
* ECOG Performance Status 0-1
* Estimated survival of ≥ 12 weeks
* Provide written informed consent

Exclusion Criteria:

* Prior chemotherapy for advanced NSCLC
* Neoadjuvant or adjuvant treatment within six (6) months of registration
* Prior radiation therapy within three (3) weeks of registration; all side effects must have resolved by registration
* Prior treatment with an investigational or marketed agent that acts by antiangiogenesis mechanisms
* Large ( > 4 cm) centrally located lesions or large lesions in close proximity to major blood vessels unless treated with palliative radiation
* Brain metastases or leptomeningeal disease, except for patients who have had a resection and/or completed a course of cranial irradiation, have no worsening CNS symptoms, and have discontinued all corticosteroids for that indication for at least one (1) month prior to registration
* History of gross hemoptysis (defined as bright red blood of at least ½ teaspoon or 2.5 mL per episode) within three (3) months of registration unless definitively treated with surgery, radiation, arteriographic embolization, or endobronchial interventions at least four (4) weeks prior to registration
* Presence of cavitory lesion
* Presence of squamous histology (mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is not acceptable)
* Peripheral neuropathy > grade 1
* Major surgery, open biopsy or significant traumatic injury within four (4) weeks of registration or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within one (1) week prior to registration
* Current, ongoing therapeutic anticoagulation with full-dose warfarin or its equivalent
* Current or recent (within ten [10] days of the first dose of study treatment) use of aspirin (at least 325 mg/day) or other NSAIDs with anti-platelet activity or treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix), or cilostazol (Pletal)
* History of prior malignancy within the past three (3) years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or treated localized prostate cancer with a current PSA of < 1.0 mg/dL on two successive evaluations, at least three (3) months apart, with the most recent evaluation no more than four (4) weeks prior to registration
* History of serious systemic disease including:

  1. Unstable angina, New York Heart Association (NYHA) ≥ Grade II or congestive heart failure
  2. Inadequately controlled hypertension (blood pressure >150/100 mmHg while taking antihypertensive medications)
  3. Unstable symptomatic arrhythmia requiring medication
  4. Myocardial infarction within six (6) months prior to registration
  5. Stroke within six (6) months prior to registration
  6. Transient ischemic attack within six (6) months prior to registration
  7. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within six (6) months prior to registration
  8. Clinically significant peripheral vascular disease or evidence of bleeding, diathesis (prone to bleeding) or coagulopathy
  9. Active systemic bacterial, fungal or viral infection, including known HCV and HIV
* Pregnancy or women who are breast-feeding; women of child-bearing potential and non-vasectomized men must agree to use effective methods of birth control during and three (3) months following treatment period and women of child-bearing potential must have a negative pregnancy test
* History of severe hypersensitivity reaction to docetaxel or any other drugs formulated with polysorbate 80
* Any other medical condition, including mental illness or substance abuse, which in the judgment of the investigator, is likely to interfere with a patient's ability to provide informed consent, cooperate, and participate in the study, or to interfere with the interpretation of the results
* Use of any investigational agent within four (4) weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of bevacizumab and pemetrexed compared to pemetrexed monotherapy during second-line treatment of Stage IIIB or IV NSCLC | Duration of study

SECONDARY OUTCOMES:
Overall Survival (OS) | Duration of the study
Objective tumor response (objective response rate [ORR]) in second-line treatment | Duration of the study
Progression-free survival (PFS) in first-line and maintenance treatment | Duration of the study
Objective tumor response (objective response rate [ORR]) in first-line and maintenance treatment | Duration of the study
Treatment safety in first-line, maintenance and second-line treatment | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P Belani, MD, Principal Investigator — Penn State Milton S. Hershey Medical Center, Penn State College of Medicine, Penn State Hershey Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Pharmatech's Active Clinical Trials — http://www.pharmatech.com/patients/find-study/